CLINICAL TRIAL: NCT02994459
Title: Adipose Tissue Glucose Uptake in Obesity (ATGD)
Brief Title: Study of Fat Tissue's Ability to Take up Sugar in the Obese Population
Acronym: ATGD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Senior Associate Dean for Research; Professor, Medicine & Nutrition; NextGen Director of Clinical and Translational Sciences Unit, University of Missouri-Columbia
Other Study IDs: 201610005
Record Dates: First submitted 2016-12-09; First posted 2016-12-15 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and adipose/muscle tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Metabolically Normal Obese (likely insulin sensitive): i) BMI ≥30.0 but <45.0 kg/m2; maximum body circumference <165 cm to ensure subjects fit into the PET/CT and MR scanners; iii) fasting blood glucose: <100 mg/dl; iv) blood glucose 2 h after an OGTT: <140 mg/dl; v) HbA1c <5.7 %; vi) fasting insulin: <20 µU/mL.
  Interventions: Other: Weight Loss
- Metabolically Abnormal Obese (likely insulin resistant): i) BMI ≥30.0 but <45.0 kg/m2; maximum body circumference <165 cm to ensure subjects fit into the PET/CT and MR scanners; iii) fasting blood glucose: ≥100 mg/dl or blood glucose 2 h after an OGTT: ≥140 or fasting insulin: >20 µU/mL.
  Interventions: Other: Weight Loss
- Metabolically Normal Lean: i) BMI ≥18.5 but <25.0 kg/m2; ii) maximum body circumference <165 cm to ensure subjects fit into the PET/CT and MR scanners; iii) fasting blood glucose: <100 mg/dl; iv) blood glucose 2 h after an OGTT: <140 mg/dl; v) HbA1c <5.7 %; vi) fasting insulin: <20 µU/mL.
- Metabolically Abnormal Lean: i) BMI ≥18.5 but <25.0 kg/m2; ii) maximum body circumference <165 cm to ensure subjects fit into the PET/CT and MR scanners; iii) iii) fasting blood glucose: ≥100 mg/dl or blood glucose 2 h after an OGTT: ≥140 or fasting insulin: >20 µU/mL.

INTERVENTIONS:
Other: Weight Loss — Diet-induced weight loss (obese only)
  Groups: Metabolically Abnormal Obese (likely insulin resistant); Metabolically Normal Obese (likely insulin sensitive)

SUMMARY:
People who are obese often have insulin resistance (inability of insulin to properly control blood sugar) and high blood sugar. However, not all people with obesity have this problem. About one-third of people with obesity have normal sugar metabolism (the way your body uses sugar). Similarly, not all people who are lean are also metabolically healthy and a subset of people who are lean are referred to as metabolically abnormal lean (MAL) or metabolically obese lean because they have the abnormalities in glucose metabolism typically associated with obesity. The reasons why some people with obesity have a problem with blood sugar control and others do not are not entirely clear. It is thought that impaired muscle sugar uptake is the main problem related to high blood sugar in people with obesity. However, adipose tissue (fat tissue) also consumes a substantial amount of blood sugar. Therefore, it is unclear whether muscle or adipose tissue (fat tissue) are primarily responsible for altered blood sugar concentrations in persons with metabolically abnormal obesity (MAO) (those with insulin resistance), compared to those with metabolically normal (healthy) obesity (MNO), or whether "healthy" adipose tissue (fat tissue) expansion in MNO people compared with lean people provides a vessel for blood sugar removal that helps maintain normal blood sugar concentration.

Accordingly, the investigators will determine the amount of sugar that is taken up by the body and in the cells of adipose tissue (fat tissue) and muscle by infusing labeled sugar into the blood and looking at its disappearance from blood and appearance in adipose tissue (fat tissue) and muscle. The investigators will also determine how well insulin, a hormone that controls blood sugar, turns on signals that stimulate sugar uptake in fat and muscle cells. These studies will be done after an overnight fast and during an infusion of sugar and insulin (hyperinsulinemic-euglycemic clamp), in sex- and age-matched people who are insulin resistant and insulin sensitive. People with obesity will also be invited to complete a ~10% diet-induced weight loss program and will be studied again after they have achieved the weight loss goal. A group of sex- and age-matched metabolically normal lean participants will serve as control group. An attempt will be made to also study a group of sex- and age-matched metabolically abnormal lean participants.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Age: greater than or equal to 18 years but <65 years
* Weight stable (i.e., ±2 kg for at least 3 months)
* Sedentary (less than 1 hour of structured exercise per week)
* No evidence of significant organ system dysfunction or disease (e.g., diabetes, impaired kidney function, cancer, etc.)

In addition, subjects must fulfill all of the following inclusion criteria.

Metabolically Normal Lean

* BMI greater than or equal to 18.5 but <25.0 kg/m2
* Fasting blood glucose: <100 mg/dl
* Blood glucose 2 h after an OGTT: <140 mg/dl
* HbA1c <5.7 %.

Metabolically Normal Obese, likely insulin sensitive

* BMI greater than or equal to 30.0 but <45.0 kg/m2
* Fasting blood glucose: <100 mg/dl
* Fasting insulin: <20 mU/l
* Blood glucose 2 h after an OGTT: <140 mg/dl
* HbA1c <5.7 %.

Metabolically Abnormal Obese, likely insulin resistant

* BMI greater than or equal to 30.0 but <45.0 kg/m2
* Fasting blood glucose ≥100 mg/dl or blood glucose 2 h after an OGTT ≥140 mg/dl or fasting insulin >20 µU/mL or HbA1c >5.7 %.

Metabolically Abnormal Lean

* BMI greater than or equal to 18.5 but <25.0 kg/m2
* Fasting blood glucose ≥100 mg/dl or blood glucose 2 h after an OGTT ≥140 mg/dl or fasting insulin >20 µU/mL or HbA1c >5.7 %.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators plan to study a total of 45 men and women of all races and ethnic groups: 15 MAO (metabolically abnormal obese, likely insulin resistant), 15 MNO (metabolically normal obese, likely insulin sensitive), and 15 lean. All three groups will be balanced with regards to sex and race/ethnicity distribution, and the two obese groups will also be matched on percent total body fat. They will also attempt to recruit 15 metabolically abnormal lean participants.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Contribution of subcutaneous adipose tissue glucose uptake to whole-body glucose disposal in people who are insulin sensitive or insulin resistant (defined as insulin-mediated glucose disposal rate) | Baseline
  Comparison of whole body and total adipose tissue glucose disposal rate assessed by using stable isotope labeled glucose tracer infusion in conjunction with dynamic PET imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators do not currently anticipate to share IPD, but will do so upon request.

REFERENCES:
- [Derived] Cao C, Koh HE, Van Vliet S, Patterson BW, Reeds DN, Laforest R, Gropler RJ, Mittendorfer B. Increased plasma fatty acid clearance, not fatty acid concentration, is associated with muscle insulin resistance in people with obesity. Metabolism. 2022 Jul;132:155216. doi: 10.1016/j.metabol.2022.155216. Epub 2022 May 13. PMID 35577100
- [Derived] van Vliet S, Koh HE, Patterson BW, Yoshino M, LaForest R, Gropler RJ, Klein S, Mittendorfer B. Obesity Is Associated With Increased Basal and Postprandial beta-Cell Insulin Secretion Even in the Absence of Insulin Resistance. Diabetes. 2020 Oct;69(10):2112-2119. doi: 10.2337/db20-0377. Epub 2020 Jul 10. PMID 32651241